CLINICAL TRIAL: NCT03348709
Title: Does Osmolality of Oral Supplements Affect Stoma Output and Natriuresis in Patients With an Ileostomy?
Brief Title: Osmolality of Oral Supplements and Ileostomy Output
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Christian Hvas, MD PhD, associate professor, University of Aarhus
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1-10-72-12-17
Record Dates: First submitted 2017-11-16; First posted 2017-11-21 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-11

CONDITIONS: Ileostomy - Stoma; Short Bowel Syndrome; Sodium Depletion; Nutritional Deficiency
MeSH Terms: conditions — Short Bowel Syndrome; Hyponatremia; Malnutrition

STUDY DESIGN:
Intervention Model Description: Double-blinded, active comparator, cross-over intervention study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomisation by Third party; Unblinded study nurse to mix and deliver study product; masking of product to ensure comparable palatability and appearance; blinding to analyses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isoosmolar (Experimental): Iso-osmolar oral supplement (276 mOsm/kg)
  Interventions: Dietary Supplement: Isoosmolar
- Hyperosmolar (Active Comparator): Hyper-osmolar oral supplement (681 mOsm/kg)
  Interventions: Dietary Supplement: Hyperosmolar

INTERVENTIONS:
Dietary Supplement: Isoosmolar — 48 hours, 800 ml per 24 hours
  Arms: Isoosmolar
Dietary Supplement: Hyperosmolar — 48 hours, 800 ml per 24 hours
  Arms: Hyperosmolar

SUMMARY:
This double-blinded, active comparator, cross-over intervention study tested the impact of two different oral supplements on ileostomy output volume and urinary sodium excretion and intestinal aquaporin expression in eight compensated patients with an ileostomy and not on home parenteral Nutrition or fluid support.

DETAILED DESCRIPTION:
Patients with an ileostomy may experience fluid and electrolyte imbalances sedondary to an unregulated intestinal loss of water and electrolytes. The osmolality of oral supplements may affect these losses. In a double-blinded, active comparator, cross-over intervention study, the investigators test the effects of substituting 800 ml of the usual fluid intake with an intake of either an isoosmolar (300 mOsm/kg) or hyperosmolar (700 mOsm/kg) supplement during 48 hours, following baseline data collection before both intervention periods. Outcome measures were stoma output volume, 24-hour urine and urinary sodium excretion, and intestinal aquaporin 3 and 8 expressions.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or more
* ilestomy established 6 weeks or more prior to inclusion
* able to drink at least 100 ml fluid per 24 hours
* i known inflammatory bowel disease, clinical remission judged by physician's global assessment (PGA)
* less than 5 kg self-reported weight change during the past 3 months

Exclusion Criteria:

* self-reported intolerance to dairy products, including lactose
* known renal insufficiency, defined by an eGFR less than 30 ml/min
* known diabetes mellitus, defined by an HbA1C > 48 mmol/mol (6.5%)
* current enteral tube feeding or parenteral fluid or Nutrition support more than twice weekly

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Stoma output | 24 hours
  24 hour stoma output weight

SECONDARY OUTCOMES:
24-hour urine production | 24 hours
  24 hour urine volume (ml)
24-hour urinary sodium excretion | 24 hours
  24-hour sodium (mmol)

CONTACTS AND LOCATIONS:
Overall Officials: Hendrik Vilstrup, Professor, Study Chair — University of Aarhus
Locations (1):
- Aarhus University Hospital, Aarhus C, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Publication of anonymised data. Data backup in accessible data platform.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: During last 6 months of study period, 10 years
Access Criteria: established researcher

REFERENCES:
- [Derived] Rud C, Pedersen AKN, Wilkens TL, Borre M, Andersen JR, Moeller HB, Dahlerup JF, Hvas CL. An iso-osmolar oral supplement increases natriuresis and does not increase stomal output in patients with an ileostomy: A randomised, double-blinded, active comparator, crossover intervention study. Clin Nutr. 2019 Oct;38(5):2079-2086. doi: 10.1016/j.clnu.2018.10.014. Epub 2018 Oct 24. PMID 30396772